CLINICAL TRIAL: NCT00775983
Title: Same-day Dilapan Versus Overnight Laminaria for Cervical Preparation for Early Second-trimester Surgical Abortion
Brief Title: Dilapan Versus Laminaria
Acronym: DvL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Eleanor Drey, MD, Associate Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1176030877
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Results first posted 2013-07-17 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-10

CONDITIONS: Cervical Preparation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laminaria (Active Comparator): laminaria placed for cervical dilation; usual standard of care in study clinic
  Interventions: Device: laminaria
- Dilapan-S (Experimental): experimental treatment
  Interventions: Device: Dilapan-S

INTERVENTIONS:
Device: laminaria — place device in cervix for dilation
  Arms: laminaria
Device: Dilapan-S — Place in cervix for dilation.
  Arms: Dilapan-S

SUMMARY:
This is a randomized, blinded clinical trial comparing overnight laminaria versus same-day Dilapan for cervical preparation for surgical abortions occurring between fourteen and eighteen weeks gestation. Comparisons will be made between procedure time, need for additional dilation, occurrence of complications, and patient and provider satisfaction.

Hypothesis:

Cervical preparation for surgical abortion, between fourteen and eighteen weeks gestation, with same-day Dilapan is non-inferior to cervical preparation with overnight laminaria within a five-minute difference.

Primary objective:

Determine differences in procedure times

Secondary objectives:

Examine complications, and need for additional dilation between early second-trimester surgical abortions performed after cervical preparation with same-day Dilapan versus those performed after cervical preparation with overnight laminaria

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy between fourteen and eighteen weeks gestation
* Request for elective abortion and certainty of decision to proceed

Exclusion Criteria:

* Incarceration
* Minor status (women younger than eighteen years)
* Allergy to Dilapan or laminaria
* Inability to speak and understand Spanish or English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Newmann SJ, Sokoloff A, Tharyil M, Illangasekare T, Steinauer JE, Drey EA. Same-day synthetic osmotic dilators compared with overnight laminaria before abortion at 14-18 weeks of gestation: a randomized controlled trial. Obstet Gynecol. 2014 Feb;123(2 Pt 1):271-278. doi: 10.1097/AOG.0000000000000080. PMID 24402587

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited for the study at the Women's Options Center at San Francisco General Hospital (SFGH) between October 2008 and February 2010. SFGH is San Francisco's county hospital and serves a diverse and mostly uninsured population.
Pre-assignment Details: Of 72 eligible and enrolled participants, 3 did not receive an abortion (2 in the Same-day Dilapan-S group, and 1 in the Overnight laminaria group).
Groups:
- Laminaria: laminaria placed for cervical dilation; usual standard of care in study clinic. The number of laminaria placed was calculated based on a predetermined formula: weeks gestational age minus ten.
- Dilapan-S: For patients between 14 0/7 and 15 6/7 weeks' gestation on the day of the abortion, 2-3 Dilapan-S were inserted. For patients between 16 0/7 and 18 0/7 weeks' gestation, 2-5 Dilapan-S were inserted. One medium laminaria was placed along with the Dilapan-S because of the theory that the laminaria would facilitate the removal of Dilapan-S before the abortion. Patients then waited four to six hours for their abortion.
Period: Overall Study
Arm/Group | Laminaria | Dilapan-S
Started | 36 | 36
Completed | 35 | 34
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Population: Of 72 eligible and enrolled participants, 3 were excluded from analysis because they did not receive an abortion (2 in the Same-day Dilapan-S group, and 1 in the Overnight laminaria group).
Groups:
- Total: Total of all reporting groups
Arm/Group | Laminaria | Dilapan-S | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 34 | 32 | 66
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24 (7) | 27 (6) | 26 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 69
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 34 | 69

OUTCOME MEASURES:

1. Primary Outcome: Procedure Time
Description: Procedure time to complete early second-trimester dilation and evacuation (D&E)
Time Frame: Day of procedure
Population: All patients who received a surgical abortion procedure were analyzed. Since three patients did not actually obtain an abortion within the study timeframe, we could not analyze their data, thus the analysis was per protocol.
Measure: Mean (Standard Error); unit: minutes
Groups:
- Overnight Laminaria: Overnight laminaria placed for cervical dilation; usual standard of care in study clinic. The number of laminaria placed was calculated based on a predetermined formula: weeks gestational age minus ten.
Arm/Group | Overnight Laminaria | Dilapan-S
Number analyzed (Participants) | 35 | 34
minutes | 5.9 (2.9) | 8.1 (5.5)
Statistical Analysis 1: Comparison: Overnight Laminaria vs Dilapan-S; Null Hypothesis: A surgical abortion performed between 14-18 weeks gestation performed after the cervix has been prepared with same-day Dilapan-S is inferior with respect to procedure time, which is specifically outside a five minute margin of non-inferiority, when compared to procedures during the same gestational duration range performed after the cervix has been prepared overnight with laminaria; Test type: Non-Inferiority or Equivalence — Power: We assumed a standard deviation of five minutes based on historical clinic data for surgical abortions during this gestational duration range, a non-inferiority margin of five minutes, and a 10% potential attrition rate to power the study for a non-inferiority hypothesis. Thirty participants in each arm gave us 95% power to conclude non-inferiority of same day Dilapan-S compared to overnight laminaria with respect to procedure time of surgical abortions between 14-18 weeks gestation; t-test, 2 sided; Mean Difference (Final Values) = 2.1, 97.5% CI 2-sided [-0.3 to 4.5]

2. Secondary Outcome: Participants Who Experienced Complications or Need for Additional Dilation
Description: Any complications, or mechanical dilation required, for early second-trimester surgical abortions performed after cervical preparation with same-day Dilapan versus those performed after cervical preparation with overnight laminaria
Time Frame: Day of procedure
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Overnight Laminaria | Dilapan-S
Number analyzed (Participants) | 35 | 34
participants
  Bleeding requiring uterotonics | 10 | 7
  Reaspiration | 2 | 3
  Cervical laceration | 1 | 0
  Additional dilation | 8 | 22

ADVERSE EVENTS:
Time Frame: Day of procedure and one-week follow-up
Description: Patients were assessed for unexpected or serious adverse events on the day of the study procedure, and were asked one week later to report any hospital or doctor visit necessitated by complications of the study procedure.
Arm/Group | Laminaria | Dilapan-S
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/34

LIMITATIONS AND CAVEATS:
-inadequate power to compare complications directly between study groups. Procedure time was chosen as a proxy for procedural difficulty and thus potential complications

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No